CLINICAL TRIAL: NCT00607022
Title: the Effects of 3 Loading Protocols on Dental Implant Stability in Healed Ridges
Brief Title: A Randomized Prospective Clinical Trial Comparing Single Tooth Implant 3 Loading Protocols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clark Stanford (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor-Investigator, Clark Stanford, Associate Dean for Research & Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 200710722
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Results first posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Dental Implant
Keywords: dental implant; early loading; traditional loading; anterior; implant stability; Subjects presenting with one tooth missing in the anterior; incisor/canine) or pre-molar regions of the mandible; or maxilla with existing teeth that were healthy; or adequately restored shall be screened.
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Intervention Model Description: This is a phase IV Post-Market evaluation of three 510K cleared implant products. One type of dental implant was used but clinically loaded with a dental crown at one of three time points, immediate at implant placement, at 6weeks or 12 weeks following implant placement. There are therefore 3 interventions being evaluated.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- immediate load (Active Comparator): immediate load of dental implant based on the bone quality determined by the insertion torque value
  Interventions: Device: dental implant
- Loading at 6 weeks (Active Comparator): delayed load (6 weeks post surgery) of dental implants based on bone quality determined by the insertion torque value
  Interventions: Device: dental implant
- Loading at 12 weeks (Active Comparator): traditional loading of dental implants (12 weeks post surgery) based on bone quality determined by the insertin torque value.
  Interventions: Device: dental implant

INTERVENTIONS:
Device: dental implant — Dental implant stability measured with the resonance frequency analyzer (Osstell, Integration Diagnostics AB, Sweden) at time of implant placement and up to 16 weeks post placement.

SUMMARY:
This is a research study to test the clinical procedure and not the FDA approved medical device. This project will screen up to 80 volunteers to enroll 40 active subjects to receive a single tooth implant on an anterior (incisor/canine) or pre-molar tooth in the mandible or maxilla (no implants will be placed in molar sites). This 3 year research study will examine the clinical effects of loading regimens on roughened surfaced implants. The proposed research project will measure the changes in mucosal healing and maturation over a three year period following implant placement. The proposed research lays the foundation for improved health care by providing surgeons and restorative dentists with data for determining the relationship between implant healing, loading pattern and bone type. The rationale that underlies the investigation is that identification of the influences of timing of load on implant stability in varying bone types will allow routine, predictable use of early loading, which, in turn, will translate into more rapid health care, and improved psychosocial well-being of the patient. If these hypotheses are correct, these results are expected to provide evidence based research data to support early loading and immediate loading of single implants in sites of adequate bone volume, and density. In addition, it is expected that these results will fundamentally advance the field of implant dentistry and bioengineering by providing information on the principles of the bone density-mechanical environment-implant stability interaction.

DETAILED DESCRIPTION:
MATERIALS AND METHODS This longitudinal human clinical trial is designed as a prospective study, to measure implant stability with the resonance frequency analyzer (Osstell, Integration Diagnostics AB, Sweden) at time of implant placement and up to 16 weeks post placement. After 16 weeks, a definitive implant abutment will be placed and a final dental crown delivered. No further follow-up will be done with the resonance frequency approach. However, all subjects will be followed through 3 years post implant placement as described for each follow-up visit. The study population consists of subjects at the University of Iowa's College of Dentistry. Subjects presenting with one tooth missing in the anterior (incisor/canine) or pre-molar regions of the mandible or maxilla with existing teeth that were healthy or adequately restored shall be screened based on the inclusion/exclusion criteria. The missing tooth is to be replaced with a fixed implant restoration on one implant.

SEQUENCE OF VISITS A. Visit 1: Screening Examination

Subjects shall be seen for evaluation and for collection of baseline data. Pre-treatment data shall be recorded on case report forms. The visit shall include:

1. Explanation to the patient of the purposes of the study and the planned procedures related to the study.
2. Explanation to the subject of the risks and possible complications of participation in the study. Patients shall be notified that inclusion in the study is for the purpose of providing implant treatment only and that no provision for other active treatments are guaranteed or implied except for care related to the implant aspect of their oral cavity. This treatment shall be agreed upon as outlined for their specific case.

Implant Site Selection: Adequate bone volume is needed to accommodate the planned endosseous dental implant. This will mean sufficient height such that the implant would not encroach on vital structures (such as inferior alveolar nerve), and sufficient width that the implant could be placed within the confines of the existing bone without dehiscence or fenestration, requiring significant grafting at time of implant placement. Typically, this will mean space dimensions will be: 6 mm or greater ridge width facial-lingual and > 6 mm in the mesial to distal dimension . If the implant can be placed and only a few screw threads are exposed, grafting is allowed to cover these threads. In the planned occlusal-gingival dimension, there must be at least 7 mm of space from the planned head of the implant to the planned occlusal plane.

The subject should be notified that inclusion in the study is conditional upon satisfying the inclusion and exclusion criteria as seen in Table 1. Only subjects satisfying the Inclusion/Exclusion criteria shall be enrolled.

The dental implant system to be used is the Astra Tech OsseoSpeed Dental Implant System (Astra Tech AB, Mölndal Sweden). This is an FDA cleared product under FDA 510k clearance act (FDA clearance 4/30/2004). This protocol calls for use of only the 4.0 mm diameter by 11 mm long dental implant (OsseoSpeed Aqua platform; Ref Number 24622; Astra Tech AB) in the anterior (incisor/canine) or posterior pre-molar regions of the mandible or maxilla. All sites must have sound natural or restored teeth/implants Mesial and Distal to the planned site of interest (Bounded Edentulous Space or BES). The patient should otherwise have a restored stable occlusion that is mutually protected. No implants will be placed in molar sites. The implant lengths accepted in the study are 11 mm. Clinical and radiographic screening will be used to limit the study to patients with sufficient bone quantity to completely encase the implant.

Upon review of the subject's health history, inclusion/exclusion criteria a screening clinical assessment will be made. Existing dental radiographs within the past 6 months shall be acceptable. No new radiographs will be made until subject enrollment and obtaining signed informed consent. The subject will be given an informed consent for the study and reviewed with the clinical study coordinator. Preliminary diagnostic impressions will made (Penta, 3M ESPE) and poured in dental stone (Whip Mix Corp., Louisville, KY). Implant subjects may have a pre-operative Cone Bean CT imaging study (Galileos; Sirona, Charlotte NC; www.sirona.com) made at the College of Dentistry's Department of Oral Maxillofacial Radiology at the discretion of the Principal Investigator following diagnostic work-up. Subjects shall be either patients of record of the College of Dentistry or shall be enrolled if new to the College. Patient records are electronic (WinDent) along with a paper version. Paper-based Case Report Forms (CRF) containing subject's medical information will be kept in one central file in a locked cabinet in the Dental Clinical Research Center. This data will be kept in a secured file accessible only by the PI and the Clinical Coordinator.

ELIGIBILITY:
Inclusion Criteria:

* The patient is 18 years or older.
* Ability to understand and sign the informed consent prior to starting the study.
* Ability and willingness to comply with all study requirements.
* Adequate oral hygiene (defined as an average Modified Sulcus Bleeding Index of 1 or less and an average Modified Plaque Index of 1 or less).
* Must be a bounded edentulous space.
* Adequate bone volume to accommodate the planned endosseous dental implant (e.g. sufficient height such that the implant would not encroach on vital structures such as inferior alveolar nerve, and sufficient width that the implant could be placed within the confines of the existing bone without dehiscence or fenestration, requiring significant grafting at time of implant placement). The only implant utilized in this protocol will be a 4.0 mm diameter by 11 mm long implant (Fixture OsseoSpeed Astra Tech).

Typically, this will mean space dimensions will be: 6 mm or greater ridge width facial-lingual and > 6 mm in the mesial to distal dimension . If the implant can be placed and only a few screw threads are exposed, grafting is allowed to cover these threads. In the planned occlusal-gingival dimension, there must be at least 7 mm of space from the planned head of the implant to the planned occlusal plane.

* Osteotome use will be allowed but there must be a minimum of 8mm of bone height from the alveolar crest to the floor of the sinus. Maximum sinus lift will be 4 mm.
* Existing teeth are healthy and adequately restored, and desired a fixed restoration on implants.
* Patient has a mutually protected occlusion.
* The patient, if of childbearing potential, had a negative pregnancy test within one week prior to surgery.

Exclusion Criteria:

* Patients who have smoked cigarettes or chewed tobacco within the past year.
* History of alcoholism or drug abuse within the past 5 years. - Severe bruxing or clenching habits
* Untreated periodontitis
* Patients at undue risk for an outpatient surgical procedure
* Presence of residual roots at the implant site- Patients with history of site development (extensive bone augmentation) at the implant site in the past 4 months.
* Placement of implant in an extraction site that had been healing for less than 2 month.
* Presence of local inflammation or mucosal diseases such as lichen planus.
* Uncontrolled diabetes (defined as HA1c > 7.0 percent).
* Current hematologic disorder or chronic use of coumarin (or similar) anti-coagulant therapies.
* History of leukocyte dysfunction and deficiencies
* Metabolic bone disorders
* History of renal failure
* History of liver disease
* Immunocompromised patients having HIV, RA, SLE or other collagen vascular disorders.
* Chronic corticosteroid use.
* Current chemotherapy
* History of use of IV-based bisphosphonates.
* History of radiation treatment to the head or neck
* Patients requiring grafting of bone or mucosal tissue at the time of implant placement which would require submersion of the implant during the healing period.
* Use of any investigational drug or device within the 30 day period immediately prior to implant surgery
* Patients requiring submersion of implants for esthetic reasons.
* Patient requiring ongoing dental treatment in the same quadrant or opposing quadrant during the initial 16 week healing period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clark Stanford, DDS, PhD, Principal Investigator — University of Iowa
Locations (1):
- The University of Iowa College of Dentistry, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Undecided
Primary data belongs to DENTSPLY-Sirona, the sponsor

RESULTS

PARTICIPANT FLOW:
Groups:
- Immediate Load: immediate load of dental implant based on the bone quality determined by the insertion torque value
  dental implant: This longitudinal human clinical trial is designed to measure implant stability with the resonance frequency analyzer (Osstell, Integration Diagnostics AB, Sweden) at time of implant placement and up to 16 weeks post placement. delivered. No further follow-up will be done with the resonance frequency approach.
- 6 Week Load: delayed load (6 weeks post surgery) of dental implants based on bone quality determined by the insertion torque value
  dental implant: This longitudinal human clinical trial is designed to measure implant stability with the resonance frequency analyzer (Osstell, Integration Diagnostics AB, Sweden) at time of implant placement and up to 16 weeks post placement. delivered. No further follow-up will be done with the resonance frequency approach.
- 12 Week Load: traditional loading of dental implants (12 weeks post surgery) based on bone quality determined by the insertin torque value.
  dental implant: This longitudinal human clinical trial is designed to measure implant stability with the resonance frequency analyzer (Osstell, Integration Diagnostics AB, Sweden) at time of implant placement and up to 16 weeks post placement. delivered. No further follow-up will be done with the resonance frequency approach.
Period: Overall Study
Arm/Group | Immediate Load | 6 Week Load | 12 Week Load
Started | 7 | 15 | 19
Completed | 6 | 15 | 19
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Load | 6 Week Load | 12 Week Load | Total
Number analyzed (Participants) | 7 | 15 | 19 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 15 | 19 | 41
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (7) | 35 (8) | 34 (5) | 34 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 10 | 25
  Male | 2 | 5 | 9 | 16
Region of Enrollment [Number; unit: participants]
  United States | 7 | 15 | 19 | 41

OUTCOME MEASURES:

1. Primary Outcome: Implant Stability Scale (ISQ) Score Change After 16 Weeks
Description: The objective of this study is to examine the change in implant stability upon three different loading regimens during the first sixteen weeks following implant placement. ISQ score (1-100), where higher score equals more stability, was assessed. The main hypotheses of the study are 1) Implant stability (ISQ) is minimally affected when physiologic load is applied to an implant during the healing process.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate Load | 6 Week Load | 12 Week Load
Number analyzed (Participants) | 7 | 15 | 19
units on a scale
  0 | 73 (6.67) | 71 (4.47) | 69 (3)
  6 weeks | 78 (2.57) | 77 (3.1) | 77 (3.0)
  12 weeks | 81 (3.3) | 81 (3.4) | 81 (3.5)
  16 weeks | 83 (3.6) | 83 (3) | 83 (2)
Statistical Analysis 1: Comparison: Immediate Load vs 6 Week Load vs 12 Week Load; Comparison between loading groups at 16 weeks - loading at baseline, Loading at 6 weeks, and loading at 12 weeks. Scores for all groups were compared at 16 weeks from implant placement; Test type: Other — Kruskal-Wallis values between each loading group and for Wilcoxon Signed Rank for measures on the mesial vs buccal side of the implant; p > 0.05, Kruskal-Wallis — 0.0501 < p < 0.9797; Kruskal-Wallis test evaluated ISQ at each time point

ADVERSE EVENTS:
Arm/Group | Immediate Load | 6 Week Load | 12 Week Load
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/15 | 0/19
Other Adverse Events (participants affected / at risk) | 0/7 | 0/15 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No